CLINICAL TRIAL: NCT00245882
Title: The Diabetes Telemonitoring (DiaTel) Study
Acronym: DiaTel
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: United States Department of Defense (U.S. Federal Agency)
Responsible Party: Frederick R. DeRubertis, MD, VA Pittsburgh Healthcare System
Organization: VA Pittsburgh Healthcare System (U.S. Federal Agency)
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 02324; 02489
Record Dates: First submitted 2005-10-27; First posted 2005-10-28 (Estimated); Last update posted 2012-09-18 (Estimated); Status verified 2012-09

CONDITIONS: Diabetes
Keywords: Telehealth; Veterans; Glycemic control; Active care management; Care coordination
MeSH Terms: conditions — Diabetes Mellitus

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Care Coordination (Active Comparator): Care Coordination with monthly follow-up by a diabetes nurse educator
  Interventions: Behavioral: Care Coordination
- Home Telemedicine (Active Comparator): Active Care Management with Home Telemedicine
  Interventions: Behavioral: Home Telemedicine

INTERVENTIONS:
Behavioral: Care Coordination — Care coordination with monthly follow-up by a diabetes nurse educator
  Other Names: Control
  Arms: Care Coordination
Behavioral: Home Telemedicine — Active care management by a nurse practitioner using home telemedicine
  Other Names: Active Care Management
  Arms: Home Telemedicine

SUMMARY:
The purpose of this research study is to compare two different methods of helping veterans with diabetes better manage their disease. This study will compare an "Active Care Management" method using home-based technology and self-monitoring techniques with a lower-intensity "Care Coordination" method based on monthly telephone contact with a nurse.

DETAILED DESCRIPTION:
The objectives of this study are to design, implement, and evaluate two medical care initiatives of different levels of intensity for veterans with diabetes and suboptimal glycemic control. The higher-intensity initiative ("Active Care Management") will use home-based technology that enables home messaging and reminders for compliance with recommended guidelines for treatment, as well as self-monitoring of blood glucose, blood pressure, and weight. Data will be transmitted to health care providers. This initiative will feature active care management, including changes in medication and/or diet implemented by the study's certified registered nurse practitioner under the supervision of a study physician in collaboration with the subject's primary care provider (PCP).

The lower-intensity initiative ("Care Coordination") will consist of care coordination in the form of monthly monitoring of subjects via telephone by the study's research nurse who will refer the subject to his/her PCP as needed for additional care. Both initiatives represent a supplementation to current usual care practices for the treatment of diabetes in the VA.

The objective of Phase Two of the study is to determine the appropriate level of subsequent management required for sustaining glycemic, blood pressure (BP), and lipid control among subjects randomized in Phase One to care coordination (CC) or to active care management (ACM). CC involved monthly telephone calls from a diabetes nurse (RN), whereas ACM involved home messaging and monitoring with the Viterion TeleHealth System plus active management of glycemia, BP, and lipids by a nurse practitioner (NP). ACM subjects transmitted blood glucose, BP, and weight measurements daily for review and intervention, if necessary, by the NP.

Subjects who complete Phase One and consent to participate in Phase Two will be randomized to subsequent management at the same or lower intensity and followed for an additional six months. Phase One ACM subjects will be randomized in Phase Two to either care coordination with monthly telephone calls (i.e., ACM-to-CC), or care coordination with monthly telephone calls plus home telehealth monitoring but with no active management by the NP (ACM-to-CCHT). CCHT subjects will continue to transmit home blood glucose, BP, and weight daily to the project office, but abnormal values will be referred to their primary care provider (PCP) for action. Phase One CC subjects will be randomized to either continued care coordination with monthly telephone calls (CC-to-CC), or referral back to their PCP for usual care (CC-to-UC). Randomization within both groups for Phase Two will be stratified according to HbA1c (<7% or >7%) at the conclusion of the subject's six-month participation in Phase One.

The primary aim of Phase Two is to assess whether glycemic, blood pressure, and lipid control at the end of an additional six months of follow-up differs for patients randomized to the four groups specified above (i.e., ACM-to-CC, ACM-to-CCHT, CC-to-CC, and CC-to-UC), adjusted for their corresponding HbA1c levels at the end of Phase One.

ELIGIBILITY:
Inclusion Criteria:

1. enrolled for primary care at a VA Pittsburgh Healthcare System (VAPHS)site with at least one visit from June 1, 2004 through December 31, 2005
2. diagnosed with diabetes mellitus with at least 12 months of ongoing pharmacologic treatment (at least one oral hypoglycemic agent, insulin, or both)
3. born in 1926 or later
4. have an HbA1c level >/= 8.0% at the last assessment (between 6/1/04 and 12/31/05)
5. have an HbA1c level >/= 7.5% (by finger stick) at the time of enrollment
6. mentally competent to give informed consent

Exclusion Criteria:

1. one or more visits to the VAPHS Diabetes Clinic from June 1, 2004 through December 31, 2005
2. metastatic or inoperable cancer
3. Child-Pugh Class B or C end-stage liver disease
4. HIV/AIDS
5. end-stage renal disease requiring dialysis
6. ongoing home oxygen therapy
7. a history of major organ transplant (i.e., heart, lung, kidney, liver)
8. residence in an institution (e.g. nursing home, personal care home, or prison)
9. incompatible telephone service (i.e., either none or digital)
10. concurrent participation in any other research protocol

Ages: 18 Years to 79 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 150 (Actual)
Dates: Start 2005-10; Primary Completion 2007-12 (Actual); Study Completion 2007-12 (Actual)

PRIMARY OUTCOMES:
HbA1c | 3 months

SECONDARY OUTCOMES:
Proportion of subjects in each cohort with HbA1c </= 7%, BP </= 130/80, LDL-cholesterol </= 100 mg/dl, and triglycerides </= 150 mg/dl at six months | 3 months, 6 months, 9 months, 12 months
Proxy measures for cost of care (number of outpatient clinic visits, emergency room visits, hospital bed days, and pharmacy costs) | 3 months, 6 months, 9 months, 12 months
For subjects not on insulin at enrollment, time to prescription of insulin | 6 months, 12 months
For subjects on insulin at enrollment, time to change in dose and/or type of insulin | 6 months, 12 months
Subject satisfaction with care | 6 months, 12 months
Factors influencing adherence to diabetes regimen | 6 months, 12 months

CONTACTS AND LOCATIONS:
Overall Officials: Frederick R DeRubertis, MD, Principal Investigator — VA Pittsburgh Healthcare System
Locations (1):
- VA Pittsburgh Healthcare System, Pittsburgh, Pennsylvania, United States

REFERENCES:
- [Derived] Stone RA, Sevick MA, Rao RH, Macpherson DS, Cheng C, Kim S, Hough LJ, DeRubertis FR. The Diabetes Telemonitoring Study Extension: an exploratory randomized comparison of alternative interventions to maintain glycemic control after withdrawal of diabetes home telemonitoring. J Am Med Inform Assoc. 2012 Nov-Dec;19(6):973-9. doi: 10.1136/amiajnl-2012-000815. Epub 2012 May 19. PMID 22610495